

## Form 01

| Centre: XXXX | Form version: 04/01/2024, Version 1.0 |
|--------------|---------------------------------------|
|--------------|---------------------------------------|

Study Number: IRAS Project ID: XXXX

Participant Identification Number for this trial:

## **CONSENT FORM**

Title of Project : Path Active; Safety and Tolerability Study. (PASTS)

Chief Investigator : Richard Leigh

To be completed by the participant

Please **INITIAL** each box

1) I confirm that I have read the information sheet dated 04.01.2024 (version 1.0) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily.

Initial

2) I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected.

Initial

3) I understand that relevant sections of my medical notes and data collected during the study may be looked at by investigators of the trial, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records (which

Initial

4) I agree that my GP can be informed of my involvement in this study.

may include them being sent a copy of this consent form).

Initial

6) I agree to take part in the above study.

Initial



| 7) I understand that the information c | | | |
|---|---|---|---|
| other research in the future, and may be shared anonymously with other researchers. | | | |
| searchers. | | | |
| | | T * | 1 |
| | | Init | .1a1 |
| 8) I would like a summary report of the | findings of this trial sent to me. | | |
| Name of patient | Signature | Date | |
| Name of person taking | Signature | Date | |
| consent (if different from researcher) | | | |
| Researcher | Signature | Date | |
| When completed: 1 form for patient, 1 to b | e kept as part of the researcher site file, | 1 to be kept | |
| with hospital notes. | | | |
| Contact details for further information | | | |

Page 2 of 2

Centre contact details